CLINICAL TRIAL: NCT07047274
Title: The Effect of Multidimensional Disaster Education on Disaster Awareness and Disaster Response Self- Efficacy Among Student Nurses Affected by the Kahramanmaraş-centered Earthquake: a Quasi- Experimental Randomized Controlled Trial
Brief Title: Disaster Education Among Student Nurses After the Kahramanmaraş Earthquake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Hanifi DÜLGER, Dr. Lecturer, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: E-23688910-050.01.04-230003832
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Earthquake; Nurses Role; Disaster Nursing
Keywords: Disaster awareness; Disaster education; Disaster response; Earthquake; Nurse candidates; Self-efficacy

STUDY DESIGN:
Intervention Model Description: 54 students were assigned to the intervention group and 54 students to the control group using the randomization method according to grade and gender strata, and the study was completed with a total of 108 students.
Who Masked: Outcomes Assessor
Masking Description: To ensure blinding, baseline and final outcome measurements were performed by a researcher other than the training investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Experimental): A web-based training program consisting of ten sessions, each lasting one hour, was implemented for the students in the intervention group. To enhance participation and reinforce learning, game-based activities related to the session topics were conducted via an online platform (Kahoot) during each session. The training content was developed based on the expert opinions of 12 professionals specializing in emergency care, public health, internal medicine, surgery, and education. Additionally, the program was structured in alignment with the emergency action plans of AFAD, the official disaster management authority in Türkiye. The training covered key topics including types and classifications of disasters, disaster awareness, risk analysis, personal protective equipment, triage, post-disaster processes, basic first aid, and the social dimensions of disasters.
  Interventions: Behavioral: Education group (DBM/BMP)
- Control Group (No Intervention): Since there were no participants with high levels of self-efficacy and awareness in the pre-test results, 54 students were randomly assigned to the control group according to gender and grade level. After the training in the intervention group was completed, the same assessment tools were re-applied to both groups and post-test data were collected. After the data were collected, the materials used in the training were shared with the control group.

INTERVENTIONS:
Behavioral: Education group (DBM/BMP) — A structured web-based training program, consisting of ten one-hour sessions, was delivered to students in the intervention group. To foster active engagement and reinforce learning outcomes, each session incorporated interactive, game-based activities through the Kahoot platform. The content of the training was developed in collaboration with a panel of 12 subject-matter experts, including specialists in emergency care, public health, internal medicine, surgery, and education. Additionally, the structure and thematic scope of the program were aligned with the emergency action guidelines of AFAD, Türkiye's official disaster management authority. The curriculum encompassed a comprehensive range of topics, including the classification of disasters, disaster awareness, risk assessment, use of personal protective equipment, triage procedures, post-disaster management, basic first aid practices, and the psychosocial dimensions of disaster response.
  Arms: Education Group

SUMMARY:
Objective: This study examines the effect of multidimensional disaster training on disaster awareness and disaster intervention self-efficacy of pre-service nurses who experienced the effects of the earthquake centred in Kahramanmaraş. Since there is not enough disaster-related training in nursing curricula, it is thought that such trainings will improve the skills of nurses. The study aims to investigate whether this training increases students' knowledge and intervention competences towards disasters.

Methods: This research is a study with a quasi-experimental design. The study was conducted with 1st and 2nd year students who were studying at a university, Department of Nursing, and had not taken public health and disaster management courses. An intervention group and a control group were formed by applying tests measuring disaster awareness and disaster response self-efficacy to the students. Web-based multidimensional disaster training consisting of 10 sessions was given to the intervention group. After the training, both groups were retested and the changes in disaster awareness and response self-efficacy were evaluated. After that, the data was analyzed with statistical tests.

DETAILED DESCRIPTION:
Disasters are events that cause widespread destruction, exceeding a society's capacity to respond without external assistance. These events may arise from natural or human-induced causes and often result in significant social and environmental consequences. Recent years have seen a marked increase in natural disasters globally. For instance, in 2022, 387 natural disasters affected 185 million people worldwide. The earthquakes that struck the Kahramanmaraş region in Turkey in February 2023 caused massive devastation, impacting over 9 million people and resulting in more than 50,000 fatalities.

To reduce disaster-related losses, integrating disaster risk planning into national policies is essential. Disaster management involves four main stages: preparedness, mitigation, response, and recovery. Among healthcare professionals, nurses have a particularly crucial role at every stage. Their awareness and response capabilities directly influence the effectiveness of disaster interventions. Therefore, strengthening nursing education in disaster preparedness is of growing importance.

Globally, disaster-related content is included in undergraduate and postgraduate nursing education, especially in high-risk areas. However, in Turkey, such content is often limited. Previous studies show that nurses' awareness and competencies in disaster response remain inadequate. While numerous studies assess nursing students' knowledge and awareness, few focus on interventions to improve disaster response self-efficacy.

This study aims to evaluate the effect of a multidimensional disaster training program on nursing students' disaster awareness and self-efficacy.

A quasi-experimental randomized controlled trial was conducted with first- and second-year nursing students who had not received prior education in public health or disaster management. From a pool of 120 eligible students, 108 were randomly assigned into intervention and control groups (54 each), based on stratification by class and gender. The sample size was calculated using G*Power software based on medium effect size assumptions.

Prior to the intervention, all participants completed a personal information form, the Disaster Response Self-Efficacy Scale (DRSES), and the Disaster Awareness Scale (DAS). As none had high initial scores, both groups were deemed suitable for the study.

The intervention group received a web-based training program consisting of ten one-hour sessions. Each session included interactive components such as Kahoot-based quizzes to enhance engagement. The curriculum was developed with input from 12 experts across various medical and educational fields and aligned with the Turkish Disaster and Emergency Management Authority's (AFAD) guidelines. Topics included types of disasters, risk analysis, use of personal protective equipment, triage, first aid, and psychosocial support.

Following the training, both groups retook the same assessments, and post-test data were collected for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Being a first- or second-year student enrolled in the Nursing Department of a university,
* Not having received any prior education related to Public Health or Disaster Management,
* Reading and approving the informed voluntary consent form and agreeing to participate in the study.

Exclusion Criteria:

* Having received prior education or training in public health, disaster preparedness, or disaster management,
* Currently enrolled in or having completed any course related to disasters, Not providing informed consent,
* Being absent during either the intervention or data collection phases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Disaster Awareness Scale (DAS) | From baseline to the end of treatment at 10 days
  Developed by Kırıkkaya and Gerdan, is a five-point Likert-type measurement tool consisting of a total of 23 items: strongly agree 5, agree 4, undecided 3, disagree 2, strongly disagree 1. The scale, which has a 5-factor structure as disaster knowledge, pre-disaster, during disaster, post-disaster and awareness of non-structural risks, has a total variance explanation level of 57%. Cronbach Alpha reliability coefficient of the scale was calculated as α=.86.
Disaster Response Self-Efficacy Scale (DRSES) | From baseline to the end of treatment 10 days
  It was developed by Hong-Yan Li. The validity and reliability studies of the Turkish form of the scale were conducted by Koca and colleagues. It consisted of 19 items and 3 sub-dimensions, and the answers were taken with a 5-point Likert scale (1=Not confident at all, 2=basically not confident, 3=Somewhat confident, 4=Basically confident, 5=Fully confident). A high score indicates a high level of disaster response self-efficacy. Cronbach's alpha coefficient of the whole scale was determined as 0.96. Cronbach alpha values for the three dimensions were determined as on-site rescue competence=0.93, psychological nursing competence in disaster=0.93 and the quality of the role undertaken in disaster and adaptation competence =0.93.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The surveys and indices used in the study can be shared by researchers.
Supporting Information: Study Protocol